CLINICAL TRIAL: NCT03514953
Title: The Impact of Physical (In)Activity on Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HM20012432
Record Dates: First submitted 2018-04-20; First posted 2018-05-03 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Sleep

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reduced Physical Activity (Experimental): Participants will reduce their physical activity level by >5000 steps per day for two weeks.
  Interventions: Behavioral: Reduced Physical Activity

INTERVENTIONS:
Behavioral: Reduced Physical Activity — Preliminary Phase (Baseline to Day 7): Subjects will begin wearing an accelerometer for 7 days to track physical activity and sleep patterns.
  Experimental Phase 1 (Day 7 to Day 21): Participants will be required to reduce their step count by 5,000 steps per day and engage in no moderate-vigorous physical activity during this timeframe. Every 7 days subjects undergo the blood draw, vascular health measures and questionnaire assessments.
  Experimental Phase 2 (Day 21 to 28): During the week of assessment, subjects will be asked to return to their normal physical activity patterns.

SUMMARY:
The proposed research will examine the role of physical activity (PA) on altering sleep quality (SQ) while systematically examining novel mechanisms that may drive changes in SQ. Specifically, the study will examine how a 2 week reduction in PA alters sleep quality in young, healthy individuals. Additionally, during this reduction in PA, the study will examine changes in inflammation, oxidative stress, and sympathetic activity to identify potential mechanisms for alterations in sleep quality.

DETAILED DESCRIPTION:
Sleep, which makes up approximately one third of an individual's life, plays a vital role in normal bodily functioning by regulating metabolic and endocrine function. Disturbed sleep, defined as any alteration to normal sleep patterns, is highly prevalent, affecting 35% and 41% of the general population in the United States and has been linked to poor cardiovascular health, diabetes, obesity, dyslipidemia, and hypertension. Young adults are a population at high risk for disturbed sleep-related health outcomes due to negative lifestyle behaviors such as alcohol consumption, drug use, study patterns, and excessive screen time that remain with advancing age. Due to the importance of improving or maintaining health outcomes through adequate sleep quality (SQ), the proposed research will examine the role of physical activity (PA) on altering SQ while systematically examining novel mechanisms that may drive changes in SQ. Specifically, this study will examine how alterations (increases and decreases) in PA impact SQ and how these alterations modify inflammation, oxidative stress, and sympathetic stimulation in young adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals with average weekly step count greater than 7500
* Low risk of cardiovascular, pulmonary, and metabolic disease

Exclusion Criteria:

* Individuals with cardiovascular, pulmonary, and metabolic disease
* Individuals taking medications that may affect cardiovascular, pulmonary, and metabolic function
* Diet differs substantially from typical diet, significant calorie restriction, or vitamin/mineral deficiencies
* Pregnant women
* Prisoners

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change in sleep quality (phase 1) | Day 7 to Day 21
  Evaluation of sleep efficiency (the ratio of total sleep time to the total time recorded in which the subject was not asleep (i.e. brief awakenings))
Change in sleep quality (phase 2) | Day 21 to Day 28
  Evaluation of sleep efficiency (the ratio of total sleep time to the total time recorded in which the subject was not asleep (i.e. brief awakenings))

SECONDARY OUTCOMES:
Level of Tumor Necrosis Factor Alpha in blood | Measured on Day 7, Day 14, Day 21, Day 28
  Measurement of inflammation with greater levels indicating more inflammation
Level of Interleukin-6 in blood | Measured on Day 7, Day 14, Day 21, Day 28
  Measurement of inflammation with greater levels indicating more inflammation
Level of Interleukin-1 in blood | Measured on Day 7, Day 14, Day 21, Day 28
  Measurement of inflammation with greater levels indicating more inflammation
Level of Norepinephrine in blood | Measured on Day 7, Day 14, Day 21, Day 28
  Measurement of catecholamine production with greater levels indicating more production
Level of Epinephrine in blood | Measured on Day 7, Day 14, Day 21, Day 28
  Measurement of catecholamine production with greater levels indicating more production
Level of Lipid peroxidation in blood | Measured on Day 7, Day 14, Day 21, Day 28
  Measurement of oxidative stress with greater levels indicating more oxidative stress
Protein oxidation in blood | Measured on Day 7, Day 14, Day 21, Day 28
  Measurement of oxidative stress with greater levels indicating more oxidative stress
Change in Lower Limb Vascular Function | Measured on Day 7, Day 14, Day 21, Day 28
  Measurement of popliteal artery dilation after 5 minutes of lower limb occlusion
Change in Upper Limb Vascular Function | Measured on Day 7, Day 14, Day 21, Day 28
  Measurement of brachial artery dilation after 5 minutes of lower limb occlusion
Change in Leg Vascular Function | Measured on Day 7, Day 14, Day 21, Day 28
  Measurement of leg blood flow during 1 minute of passive leg movement

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Garten, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States